CLINICAL TRIAL: NCT07039929
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Multiple-Dose, Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of INCB000631 When Administered Orally to Healthy Adult Participants
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of INCB000631 When Administered Orally to Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Business Decision
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INCB000631-102
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Healthy Participants
Keywords: INCB000631

STUDY DESIGN:
Intervention Model Description: Cohorts C and D will be dosed either once daily (Treatment A) or twice daily (Treatment B) not both.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort A (Experimental): INCB000631 or placebo will be administered at the protocol defined dose based on cohort assignment.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort B (Experimental): INCB000631 or placebo will be administered at the protocol defined dose based on cohort assignment.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort C Treatment A (Experimental): INCB000631 or placebo will be administered at the protocol defined dose based on cohort assignment.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort C Treatment B (Experimental): INCB000631 or placebo will be administered at the protocol defined dose based on cohort assignment.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort D Treatment A (Experimental): INCB000631 or placebo will be administered at the protocol defined dose based on cohort assignment.
  Interventions: Drug: INCB000631; Drug: Placebo
- Cohort D Treatment B (Experimental): INCB000631 or placebo will be administered at the protocol defined dose based on cohort assignment.
  Interventions: Drug: INCB000631; Drug: Placebo

INTERVENTIONS:
Drug: INCB000631 — Oral; Tablet
Drug: Placebo — Oral; Tablet

SUMMARY:
This study will be conducted to assess the safety, tolerability, and pharmacokinetics of INCB000631 when administered orally to healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Age 19 to 55 years (in compliance with Nebraska state law), inclusive, at the time of signing the ICF.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at screening.
* No clinically significant findings on screening evaluations (clinical, laboratory [except lipids], and ECG).
* Ability to swallow and retain oral tablets.
* Willingness to avoid pregnancy or fathering children based on the criteria below.

  * Male participants with reproductive potential must agree to take appropriate precautions to avoid fathering children, including refraining from donating sperm, from screening through 90 days (a spermatogenesis cycle) after the last dose of study drug. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * All female participants must have a negative pregnancy test at screening and a negative pregnancy test at check-in (Day -1) and must agree to take appropriate precautions to avoid pregnancy and refrain from donating oocytes from screening through 30 days (1 menstrual cycle) after the last dose of study drug. Permitted methods in preventing pregnancy should be communicated to the participants and their understanding confirmed.
  * Female participants not considered to be of childbearing potential as defined in the protocol are eligible and must have a negative pregnancy test at screening and check-in.

Exclusion Criteria:

* History of uncontrolled or unstable respiratory, renal, gastrointestinal, endocrine, pulmonary, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening.
* History of an autoimmune disease (eg, myasthenia gravis).
* History of cardiovascular, cerebrovascular, cerebral, peripheral vascular, or thrombotic disease or uncontrolled hypertension.
* High blood pressure (systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mm Hg at screening, confirmed by repeat testing).
* Confirmed resting pulse (up to 3 measurements) < 40 bpm or > 100 bpm at screening for vital signs.
* History or presence of an abnormal ECG before initial dose administration.
* Presence or history of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn disease or chronic pancreatitis).
* History of malignancy within 5 years of screening, with the exception of cured basal cell or squamous cell carcinoma of the skin, ductal carcinoma in situ, or Gleason 6 prostate cancer.
* History of other malignancy within 2 years of screening (with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy) or cancers from which the participant has been disease-free for < 1 year after treatment with curative intent.
* Current or recent (within 3 months of screening) clinically significant gastrointestinal disease or surgery (including cholecystectomy; excluding appendectomy and hernia repair) that could affect the absorption of study drug.
* Hemoglobin, WBC count, platelet count, or absolute neutrophil count less than the laboratory lower limit of normal at screening or at check-in, confirmed by repeat testing (up to twice).
* Hepatic transaminases (ALT and AST), ALP, or total bilirubin > 1.25 × the laboratory-defined ULN.
* Any major surgery within 4 weeks of screening.
* Donation of blood to a blood bank or participation in a clinical study (except a screening visit) within 4 weeks of screening (within 2 weeks for donation of plasma only).
* Blood transfusion within 4 months of check-in (Day -1).
* Chronic, known, or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment (includes latent tuberculosis).
* Positive test for HBV, HCV, or HIV.
* Receipt of any vaccine (including attenuated) within 3 months of the planned start of the study drug or anticipation of need for such a vaccine during the study. This includes seasonal influenza vaccines.
* History of significant alcohol use within 3 months of screening, defined as regular alcohol consumption > 21 units per week for males and > 14 units for females (1 unit = one-half pint of beer or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine).
* Positive urine or breath test for ethanol or positive urine or serum screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Consuming alcoholic beverages from 7 days before check-in until discharge from the CRU.
* Ingestion of caffeine- or xanthine-containing products (eg, coffee, tea, cola drinks, energy drinks, and chocolate) within 48 hours before check-in until after collection of the final PK and/or PD sample.
* Consumption of Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices within 48 hours before check-in.
* Using nicotine-containing products 7 days before check-in until after discharge from the CRU.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with another investigational medication or current enrollment in another investigational drug study.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with an inducer or inhibitor of CYP3A4, P-gp, or BCRP.
* Current use of prohibited medication.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity).
* Inability to undergo venipuncture or tolerate venous access (participant has inadequate veins for repeat venipuncture or venous access.
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations.
* Use of prescription drugs (including hormonal contraceptives) within 14 days of study drug administration or nonprescription medications/products (including minerals and phytotherapeutics/herbals [including St John's wort]/plant-derived preparations) within 7 days of study drug administration. However, occasional and standard-dose acetaminophen and standard-dose vitamins are permitted. Megadose vitamins or supplements are not permissible.
* Pregnant or breastfeeding.
* Excessive exercise beyond the activities of daily living (eg, triathlon/biathlon, marathons) within 7 days before check-in (Day -1).

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2025-07-28 (Actual); Primary Completion 2025-10-11 (Actual); Study Completion 2025-10-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2.5 months
  Defined as any adverse event, either reported for the first time or the worsening of a pre-existing event, occurring after dose of study drug.
PK for plasma INCB000631: Cmax | Up to Day 18
  Maximum Observed Plasma Concentration of INCB000631.
PK for plasma INCB000631: tmax | Up to Day 18
  Time to maximum plasma concentration of INCB000631.
PK for plasma INCB000631: AUC(0-12) | Up to Day 18
  Area under the plasma concentration-time curve from Hour 0 to 12.
PK for plasma INCB000631: AUC(0-24) | Up to Day 18
  Area under the plasma concentration-time curve from Hour 0 to 24.
PK for plasma INCB000631: Ctrough | Up to Day 18
  Observed plasma concentration before the next dose of INCB000631.
PK for plasma INCB000631: AUCτ | Up to Day 18
  Area under the plasma concentration-time curve during the dosing period "τ".
PK for plasma INCB000631: AUC∞ | Up to Day 18
  Area under the plasma concentration-time curve from time t to infinity.
PK for plasma INCB000631: AUClast | Up to Day 18
  Area under the plasma concentration-time curve to the last time point.

SECONDARY OUTCOMES:
PK for plasma INCB000631: t1/2 | Up to Day 18
  Apparent terminal phase disposition half-life of INCB000631.
PK for plasma INCB000631: CL/F | Up to Day 18
  Dose clearance of INCB000631.
PK for plasma INCB000631: Vz/F | Up to Day 18
  Apparent oral dose volume of distribution of INCB000631.
PK for plasma INCB000631: λz | Up to Day 18
  Apparent terminal-phase disposition rate constant of INCB000631.
PK for urine INCB000631: Ae | Up to Day 18
  Amount of INCB000631 excreted in the urine over sampling interval.
PK for urine INCB000631: Ae24h | Up to Day 18
  Amount of INCB000631 excreted in the urine over 24 hours.
PK for urine INCB000631: Ae360h | Up to Day 18
  Amount of INCB000631 excreted in the urine over 360 hours.
PK for urine INCB000631: fe | Up to Day 18
  Percent of INCB000631 excreted in the urine.
PK for urine INCB000631: CLR | Up to Day 18
  Renal clearance of INCB000631.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Celerion, Inc, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study to Assess the Safety, Tolerability, and Pharmacokinetics of INCB000631 When Administered Orally to Healthy Adult Participants — https://www.incyteclinicaltrials.com/trials/INCB000631-102